CLINICAL TRIAL: NCT03443388
Title: A Pilot Study of the Safety of a Novel Helmet Design in Patients With Seizures
Brief Title: Novel Helmet Design in Patients With Seizures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael A. Gelfand, MD, PhD (Other)
Collaborators: Epilepsy Foundation (Other)
Responsible Party: Sponsor-Investigator, Michael A. Gelfand, MD, PhD, Assistant Professor of Clinical Neurology, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 824620
Record Dates: First submitted 2018-02-07; First posted 2018-02-23 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Drug Resistant Epilepsy; Drop Seizures; Generalized Tonic Clonic Seizure; Complex Partial Seizure; Fall Due to Seizure
Keywords: head injury from seizures; seizures resulting in fall; helmet for seizures; novel helmet design; inflatable helmet; Hovding Inc; helmet; device
MeSH Terms: conditions — Drug Resistant Epilepsy; Syncope; Epilepsy, Tonic-Clonic; Seizures

STUDY DESIGN:
Intervention Model Description: This is an open-label, randomized, 2-way crossover pilot safety study of the Hövding helmet device in patients with drug resistant epilepsy. Reference therapy is no head-protective device. Part 1 will test helmets on 4 normal controls falling from standing. If the helmet deploys in at least 3 out of 4 falls, we will proceed to Part 2. Part 2 will enroll up to 20 patients with Drug Resistant Epilepsy. Patients will be block randomized to first wear the helmet in their daily lives until helmet deployment or for up to 3 months, or to first not wear a helmet for up to 3 months. Patients in each group will complete self-administered questionnaires. We will compare circumstances, injuries, and post concussive scales in seizures resulting in falls occurring while the helmet was worn versus seizures resulting in falls occurring while the helmet was not being worn using daily seizure calendar, medical records review, the Rivermead Post Concussive Scale and other qualitative questionnaires.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Part 2: Helmet (Active Comparator): After a screening period, 10 patients with drug resistant epilepsy will first be assigned to wear one Hövding inflatable helmet in their daily lives. Subjects will fill out questionnaires about their seizures, injuries, and the circumstances of inflation when it occurs. After experiencing a seizure resulting in a fall or any helmet deployment, patients will crossover to the "no helmet" group. If no seizure resulting in fall occurs in 3 months, participation will end.
  Interventions: Device: Hövding inflatable helmet
- Part 2: No Helmet (No Intervention): After a screening period, 10 subjects with drug resistant epilepsy will first be assigned to not wear an inflatable helmet. Subjects will fill out questionnaires about their seizures and injuries. After approximately 3 months, patients will crossover to the "helmet" group.

INTERVENTIONS:
Device: Hövding inflatable helmet — The Hövding inflatable helmet is designed for cyclists as a collar with a deployable airbag that inflates when a sensor detects rapid changes in acceleration. The inflated helmet wraps the back and sides of the user's head in inflated nylon fabric which then slowly deflates after deploying.
  Arms: Part 2: Helmet

SUMMARY:
This is a two-part study that aims to determine the reliability and safety of the use of the Hövding inflatable helmet in seizures, as evidenced by the deployment of the helmet during seizures, and qualitative patient reporting.

DETAILED DESCRIPTION:
Part 1: 4 healthy volunteers will fall from a standing position onto a padded surface to evaluate for consistent helmet deployment from a standing position. Part 2: up to 20 patients with drug resistant epilepsy who do not use existing head-protective devices will be enrolled and assigned to first enter "helmet" or "no helmet" groups. When assigned to the "helmet" group, patients will wear the helmet until deployment during a seizure or up to 3 months. Subjects will complete questionnaires about their seizures including any injuries sustained, post concussive symptom questionnaire, and the circumstances of inflation. Patients will return to site after helmet deployment. While assigned to the "no helmet" group, patients will complete the same questionnaires, except those relating to helmet inflation. We will compare circumstances, injuries, and post concussive scales in seizures resulting in falls occurring while the helmet was worn versus seizures resulting in falls occurring while the helmet was not being worn.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

1. Age 18-60 at the time of enrollment.
2. Have neck circumference between 34 and 42 cm.
3. Can understand and provide written informed consent.
4. Must be competent to follow all study procedures.
5. Able to read, speak, and understand English.

Part 2:

1. Have at least one seizure every 6 months that might result in a fall (Generalized Tonic Clonic Seizure, Atonic Seizure, and/or Complex Partial Seizure resulting in a fall).
2. Has a seizure frequency of at least once per 2 months.
3. Be between ages 18-65 at the time of enrollment.
4. Have neck circumference between 34 and 42 cm
5. Must live in a home with electrical power supply.
6. If female and of childbearing potential, has negative pregnancy test at the beginning of the study and willing to use appropriate birth control for the duration of the study.
7. Can understand and sign written informed consent.
8. Must be competent to follow all study procedures.
9. Able to read, speak, and understand English.

Exclusion Criteria:

Part 1:

1. Subject is currently pregnant

Part 2:

1. Patient already wears a helmet for seizure safety.
2. Subject is pregnant, planning to become pregnant during the study, or is unwilling to use an appropriate form of birth control during the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2020-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gelfand, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
Hövding Inc. may receive the used helmets and the information about how they were deployed. All information shared will be deidentified.

REFERENCES:
- [Background] King NS, Crawford S, Wenden FJ, Moss NE, Wade DT. The Rivermead Post Concussion Symptoms Questionnaire: a measure of symptoms commonly experienced after head injury and its reliability. J Neurol. 1995 Sep;242(9):587-92. doi: 10.1007/BF00868811. PMID 8551320

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4 subjects for part 1. 5 subjects for part 2
Groups:
- Part 1: Staged Fall: Four healthy volunteers were enrolled in Phase 1 of the study to assess the reliability of helmet deployment during staged falls
- Part 2: Helmet First, Then no Helmet; Part 2: No Helmet First, Then Helmet: This was a randomized crossover study; subjects were initially randomized to either 'helmet' or 'no helmet' groups; after the first evaluable fall they crossed into the other group.
Period: Overall Study
Arm/Group | Part 1: Staged Fall | Part 2: Helmet First, Then no Helmet | Part 2: No Helmet First, Then Helmet
Started | 4 | 3 | 2
Completed | 4 | 2 | 2
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 2 (Crossover): All participants who agreed to participate in Phase 2 of the study
- Phase 1 (Staged Fall): All participants who agreed to participate in Phase 1 of the study
- Total: Total of all reporting groups
Arm/Group | Phase 2 (Crossover) | Phase 1 (Staged Fall) | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 39 [26 to 54] | 36.5 [27 to 44] | 39 [26 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 3 | 2 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 9
Type of Epilepsy [Count of Participants; unit: Participants]
  Focal Epilepsy | 3 | 0 | 3
  Generalized Epilepsy | 1 | 0 | 1
  Lennox-Gastaut Syndrome | 1 | 0 | 1
  No epilepsy diagnosis (control) | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Successful Deployments
Description: 3 out of 4 successful deployments was set as a criteria to allow advancement to part 2.
Time Frame: 1 day
Measure: Number; unit: number of successful deployments
Units Other Than Participants: Helmet Deployments
Groups:
- Phase 1: Staged Fall: Participants with a singular staged fall
Arm/Group | Phase 1: Staged Fall
Number analyzed (Participants) | 4
Number analyzed (Helmet Deployments) | 4
number of successful deployments
  Successful Helmet Deployments | 4
  Unsuccessful Helmet Deployments | 0

2. Primary Outcome: Part 2: Helmet Deployment Questionnaire
Description: Differences in Helmet Deployment Questionnaire responses will be compared between subjects wearing helmets during a seizure, and subjects not wearing helmets during a seizure.
Time Frame: 6 months
Population: 3 participants had evaluable falls with the helmet; 2 participants had evaluable falls without a helmet. Only 1 patient had an evaluable fall in both helmet and no-helmet conditions.
Measure: Number; unit: participants
Groups:
- Helmet: Participants randomized to helmet
- No Helmet: Participants randomized to no helmet
Arm/Group | Helmet | No Helmet
Number analyzed (Participants) | 5 | 5
participants
  Participants with evaluable falls | 3 | 2
  Participants without evaluable fall | 2 | 2
  Participants lost to follow up before evaluation of fall completed | 0 | 1
  Helmet did not deploy with evaluable fall: number analyzed (Participants) | 3 | 0
  Helmet did not deploy with evaluable fall | 1 |
  helmet deployed after evaluable fall: number analyzed (Participants) | 3 | 0
  helmet deployed after evaluable fall | 2 |
  Patients with Minor Abrasions/Lacerations to head after a fall: number analyzed (Participants) | 3 | 2
  Patients with Minor Abrasions/Lacerations to head after a fall | 0 | 2
  Patients with ER visit due to fall: number analyzed (Participants) | 3 | 2
  Patients with ER visit due to fall | 0 | 1

3. Secondary Outcome: Rivermead Post Concussive Scale
Description: Differences in head injury symptoms as reported using the Rivermead Post Concussive Scale will be compared between subjects wearing helmets during a seizure, and subjects not wearing helmets during a seizure, and also between subjects following a seizure in which the helmet deployed, and seizures in which the helmet was either not being worn or did not deploy. The scale for each item of this survey: 0 = not experienced at all 1 = no more of a problem 2 = a mild problem 3 = a moderate problem 4 = a severe problem. Each item was assessed as "compared with before the accident, do you now (i.e., over the last 24 hours) suffer from:" or "Are you experiencing any other difficulties?" with a write in option with the same scale. A lower score on each item is better, indicating lesser symptom severity compared to prior to falling with or without the helmet. The score for each item is summed to obtain each patient's total, indicative of total symptom severity. Total range from 0 - 72.
Time Frame: 6 months
Population: Rivermead scales were not collected consistently enough to be analyzed as intended. However, data presented include average Rivermead score of those for whom data was obtained. No individual participant completed the scale at each time point. Data was obtained for one participant with a fall with helmet (0, helmet did not deploy), and two participants with a fall without a helmet (0 and 43).
Measure: Mean (Full Range); unit: Average Rivermead Score
Groups:
- Phase 2 Participant Data: Participants randomized to helmet
- Participants Randomized to no Helmet: Participants who
Arm/Group | Phase 2 Participant Data | Participants Randomized to no Helmet
Number analyzed (Participants) | 1 | 2
Average Rivermead Score | 0 [0 to 0] | 21.5 [0 to 43]

4. Secondary Outcome: Seizure Questionnaire
Description: Differences in Seizure Questionnaire responses detailing circumstances of seizure and any injuries sustained will be compared between subjects wearing helmets during a seizure, and subjects not wearing helmets during a seizure, and also between subjects following a seizure in which the helmet deployed, and seizures in which the helmet was either not being worn or did not deploy.
Time Frame: 6 months
Population: Participants who were or did not wear the helmet for whom data is available (e.g., were not lost to follow up).
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2 Participants Who Wore the Helmet: Participants who wore the helmet
- Phase 2 Participants Not Wearing Helmet: Participants who did not wear helmet
Arm/Group | Phase 2 Participants Who Wore the Helmet | Phase 2 Participants Not Wearing Helmet
Number analyzed (Participants) | 5 | 4
Participants
  Injury resulting from evaluable fall | 0 | 2
  No injury resulting from fall | 3 | 0
  No evaluable fall | 2 | 2

5. Secondary Outcome: Injury-related Medical Record Review
Description: Differences in injuries resulting from a seizure per injury-related medical record review will be compared between subjects wearing helmets during a seizure, and subjects not wearing helmets during a seizure, and also between subjects following a seizure in which the helmet deployed, and seizures in which the helmet was either not being worn or did not deploy.
Time Frame: 6 months
Population: No individual subject had falls from seizures during both the helmet and no-helmet periods.
Measure: Count of Participants; unit: Participants
Groups:
- Helmet: Participants in phase 2 who wore the helmet
- No Helmet: Participants in phase 2 who did not wear the helmet
Arm/Group | Helmet | No Helmet
Number analyzed (Participants) | 5 | 4
Participants
  Participants who had an evaluable fall | 3 | 2
  Participants who had an evaluable fall caused by a seizure: number analyzed (Participants) | 3 | 2
  Participants who had an evaluable fall caused by a seizure | 1 | 2
  Participants whose helmet deployed during a non-seizure evaluable fall: number analyzed (Participants) | 3 | 0
  Participants whose helmet deployed during a non-seizure evaluable fall | 2 |
  Participants whose helmet did not deploy during an evaluable fall: number analyzed (Participants) | 3 | 0
  Participants whose helmet did not deploy during an evaluable fall | 1 |
  Participants injured after evaluable fall: number analyzed (Participants) | 5 | 2
  Participants injured after evaluable fall | 0 | 2

6. Secondary Outcome: Helmet Deployment Questionnaire (Seizure/Not Seizure)
Description: Differences in helmet deployment questionnaire responses describing events of helmet deployment during seizures resulting in falls will be compared with responses describing helmet deployment (per day of use) not associated with seizure.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Helmet: Participants who experienced an evaluable fall while wearing helmet
Arm/Group | Helmet
Number analyzed (Participants) | 3
Participants
  Helmet deployed during fall from seizure | 0
  Helmet did not deploy | 0
  Helmet deployed when standing while having a seizure | 1
  Helmet deployed for a non-seizure related fall | 1
  Helmet deployed while sitting rapidly from standing | 1

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Phase 1: All participants in phase 1
- Phase 2: Subjects Wearing a Helmet: All participants in phase 2 who wore a helmet
- Phase 2: Subjects Not Wearing a Helmet: All participants randomized in phase 2 who did not wear a helmet
Arm/Group | Phase 1 | Phase 2: Subjects Wearing a Helmet | Phase 2: Subjects Not Wearing a Helmet
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5 | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 (N=4) | Phase 2: Subjects Wearing a Helmet (N=5) | Phase 2: Subjects Not Wearing a Helmet (N=4)
Minor abrasions/head lacerations (Musculoskeletal and connective tissue disorders) | NA | NA | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/88/NCT03443388/Prot_SAP_001.pdf